CLINICAL TRIAL: NCT03373877
Title: A Phase Ib Study of Ruxolitinib in Combination With PU-H71 for the Treatment of Subjects With Primary Myelofibrosis (PMF), Post-Polycythemia Vera MF (Post-PV MF), and Post-EssentialThrombocythemia MF (Post-ET MF)
Brief Title: Evaluation of Ruxolitinib in Combination With PU-H71 for Treatment of Myelofibrosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Samus is focusing all of their efforts in myelofibrosis on the new oral formulation of PU-H71.
Sponsor: Samus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PU-H71-01-002
Record Dates: First submitted 2017-11-29; First posted 2017-12-14 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Myelofibrosis; Primary Myelofibrosis; Post-polycythemia Vera Myelofibrosis; Post-essential Thrombocythemia Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — 9H-purine-9-propanamine, 6-amino-8-((6-iodo-1,3-benzodioxol-5-yl)thio)-N-(1-methylethyl)-; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose 1: PU-H71 225 mg/m2 + ruxolitinib (Experimental): Cohort 1
  Interventions: Drug: PU-H71; Drug: Ruxolitinib
- Dose 2: PU-H71 300 mg/m2 + ruxolitinib (Experimental): Cohort 2
  Interventions: Drug: PU-H71; Drug: Ruxolitinib
- Dose 3: PU-H71 400 mg/m2 + ruxolitinib (Experimental): Cohort 3
  Interventions: Drug: PU-H71; Drug: Ruxolitinib
- Dose 4: PU-H71 600 mg/m2 + ruxolitinib (Experimental): Cohort 4
  Interventions: Drug: PU-H71; Drug: Ruxolitinib

INTERVENTIONS:
Drug: PU-H71 — PU-H71 treatments will be administered by IV infusion on days 1, 8, and 15 of each 28-day cycle.
Drug: Ruxolitinib — Dosing will be in accordance with current package insert and dose subject was on during study entry.
  Other Names: Jakafi

SUMMARY:
This is a multicenter 2-part, Phase 1b study designed to assess the safety, tolerability, pharmacokinetics (PK) and preliminary efficacy of PU-H71 in subjects taking concomitant ruxolitinib. The first part (Dose Escalation) will employ a standard 3+3 dose escalation design to determine Maximum Tolerated Dose (MTD). The second part of the study (Dose Confirmation) will confirm the recommended Phase 2 dose (RP2D) in an expanded population.

DETAILED DESCRIPTION:
This is a multicenter 2-part, Phase 1b study designed to assess the safety, tolerability, PK and preliminary efficacy of PU-H71 (dihydrochloride salt) in subjects taking concomitant ruxolitinib. The first part (Dose Escalation) will employ a standard 3+3 dose escalation design to determine MTD. The second part of the study (Dose Confirmation) will confirm the RP2D in an expanded population.

Up to 30 subjects who have active disease despite having received a minimum of 6 months of ruxolitinib therapy (including last 2 months at a daily dose of ≥5 mg twice daily and no more than one dose reduction 2-8 weeks prior to the baseline visit)stable dose will be enrolled to evaluate the safety, PK, and MTD of IV PU-H71 administered in combination ruxolitinib. Four ascending dose levels are planned. The planned dose levels of PU-H71 are 225 mg/m2, 300 mg/m2, 400 mg/m2, and 600 mg/m2. Additional dosing cohorts may be added at the discretion of the Safety Review Committee (SRC).

Following a 28-day screening period, eligible subjects will receive PU-H71 once weekly intravenously for three consecutive weeks, followed by one week off on a 28-day cycle (D1, D8, D15, every 28 days). Ruxolitinib will be administered twice daily per the package insert at the stable dose the subject had been receiving prior to enrolling in the study.

Subjects will have pk samples taken and ECGs performed at various time points throughout the study. Subjects will have safety evaluations including physical examinations, vital signs, laboratory assessments, and AE reporting. If deemed necessary, additional safety measurements will be performed at the discretion of the Investigator or the SRC.

Subjects will be treated until disease progression, DLT, death, or study termination.

At each dose level, a 3+3 dose escalation design will be employed. If none of the initial 3 subjects in the cohort experience a DLT within the first cycle, a new cohort of 3 subjects will be treated at the next higher dose level. If 1 of the 3 subjects in a cohort experiences a DLT, then 3 additional subjects will be treated at the same dose level as described under Dose Limiting Toxicities.

Once the MTD has been determined in the dose escalation portion of the study, up to 15 patients may be enrolled for further evaluation of safety, PK, and preliminary clinical activity in a dose confirmation phase.

A safety review committee (SRC) will assess the safety, tolerability, and available PK information collected for each dose level, decide whether to proceed to the next cohort, and determine the dose for the cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has a confirmed diagnosis of myelofibrosis, including PMF, post-PV MF, and post-ET MF.
2. Subject has been receiving ruxolitinib therapy for intermediate or high-risk myelofibrosis for >6 months prior to enrollment with no more than 1 dose reduction of ruxolitinib in the 2-8 weeks prior to enrollment and a stable daily dose ≥5 mg twice daily (BID) >2 months prior to enrollment.
3. Subject has MF with evidence of persistent disease despite ruxolitinib monotherapy treatment, consisting of:

   1. Persistent or worsening disease-related symptoms, including but not limited to fatigue, pruritus, night sweats, early satiety, and other symptoms as determined by a MPN-SAF TSS score of >20 points; AND
   2. Documented splenomegaly of at least 5 cm below the costal margin as measured on inspiration by physical exam.
4. Subject has an Eastern Cooperative Oncology Group performance status of 0-2.
5. Acceptable pre-study organ function during screening defined as:

   1. Absolute neutrophil count (ANC) ≥ 1000/uL
   2. Hemoglobin (hgb) ≥ 8.0 g/dL (may be supported with transfusion)
   3. Platelets (plt) ≥ 75,000/uL
   4. AST/SGOT and ALT/SGPT ≤2 x Upper Limit of Normal (ULN)
   5. Direct serum bilirubin ≤ 1.5 x ULN
   6. Creatinine clearance >50 mL/min/1.73 m2 based on Cockcroft Gault equation.

Exclusion Criteria:

1. Subject has known active liver disease, including viral hepatitis or cirrhosis.
2. Subject has known or suspected HIV or other active infections requiring acute or chronic treatment with systemic antibiotics. Conditions requiring topical antibiotics are acceptable.
3. Subject has a QTcF > 480 ms (corrected) in the screening or baseline ECG.
4. Subject has left ventricular ejection fraction (LVEF) ≤ 50%, or below institution's lower limit of normal (whichever is lower) by echocardiogram (ECHO) or multigated acquisition (MUGA) scan.
5. Subject has a history (or family history) of long QT syndrome.
6. Subject has coronary artery disease with an ischemic event within 6 months prior to enrollment.
7. Subject has a permanent cardiac pacemaker.
8. Subject has history of a second primary malignancy within the past 2 year except for the following (if appropriately treated and considered cured): stage I endometrial, surgically treated cervical or prostate carcinoma, and non-melanoma skin cancer.
9. Subject has significant uncontrolled medical condition within 6 months prior to enrollment, as determined by the investigator.
10. Subject has concurrent participation in any interventional studies within 14 days of first dose of study drug.
11. Subject has uncontrolled diabetes mellitus, in the judgment of the Principal Investigator.
12. Subject has an active ocular condition that in the opinion of the investigator may alter visual acuity during the course of the study (i.e., ocular inflammatory disease etc.) or a history or anticipation of major ocular surgery (including cataract extraction, intraocular surgery, etc.) during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2019-10-17 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | 12 months
  Safety of PU-H71 in combination with ruxolitinib as assessed by the incidence and severity of adverse events (AEs) and serious AEs as determined by the NCI CTCAE v4.03.
Maximum Tolerated Dose of PU-H71 (MTD) | 7 months
  MTD as assessed by the occurrences of dose limiting toxicities of PU-H71 in combination with ruxolitinib. The MTD will be defined as the dose that does not exceed an acceptable threshold of toxicity.
Recommended Phase 2 Dose of PU-H71 (RP2D) | 12 months
  The RP2D is the dose with an acceptable risk/benefit ratio that warrant study in future trials
Pharmacokinetic profile of PU-H71: Area under the plasma concentration versus time curve (AUC) | 12 months
  Area under the plasma concentration versus time curve (AUC)
Pharmacokinetic profile of PU-H71: Trough plasma concentration (Cmin) | 12 months
  Trough plasma concentration (Cmin)
Pharmacokinetic profile of PU-H71: Peak plasma concentration (Cmax) | 12 months
  Peak plasma concentration (Cmax)
Pharmacokinetic profile of PU-H71: Time to maximum plasma concentration (Tmax) | 12 months
  Time to maximum plasma concentration (Tmax)
Pharmacokinetic profile of PU-H71: Plasma half-life (T1/2) | 12 months
  Plasma half-life (T1/2)

SECONDARY OUTCOMES:
Treatment Response | 12 months
  Treatment response is to be evaluated using the revised IWG-MRT response criteria.
Symptom Burden Assessment | 12 months
  The symptomatic burden will be serially evaluated using the MPN-SAF TSS.
Biological Markers | 12 months
  Assess the effects of treatment on biological markers of the disease (i.e., bone marrow histology; JAK2V617F, CALR, or MPLW515L/K allele burden; cytogenetic response; serum cytokine profiles; and other biomarkers of disease activity).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Morgan, MS, JD, Study Director — Sponsor GmbH
Locations (10):
- United States (10):
  - Yale Cancer Center, New Haven, Connecticut
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic - Taussig Cancer Institute, Cleveland, Ohio
  - Abramson Cancer Center - University of Pennsylvania, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Mays Cancer Center UT Health San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No